CLINICAL TRIAL: NCT06904196
Title: Lenvatinib Combined With Yttrium-90 Selective Internal Radiation Therapy (SIRT) Versus Lenvatinib Alone in TACE-Refractory Hepatocellular Carcinoma: A Prospective Non-Randomized Controlled Study
Brief Title: Lenvatinib Plus SIRT vs Lenvatinib in TACE-Refractory HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIIR-21
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: hepatocellular carcinoma; Lenvatinib; Yttrium-90
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; Sirtuins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Len+SIRT (Experimental): Lenvatinib plus SIRT
  Interventions: Combination Product: Lenvatinib plus SIRT
- LEN (Active Comparator): Lenvatinib alone
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Combination Product: Lenvatinib plus SIRT — Lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. QD will be started at 3-7 days after the first SIRT.
  Arms: Len+SIRT
Drug: Lenvatinib — Lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. QD.
  Arms: LEN

SUMMARY:
This study is conducted to evaluate the efficacy and safety of lenvatinib plus SIRT (LEN+SIRT) compared with lenvatinib (LEN) alone for patients with hepatocellular carcinoma (HCC) refractory to transarterial chemoembolization (TACE).

DETAILED DESCRIPTION:
This is a prospective, non-randomized controlled trial to evaluate the efficacy and safety of LEN+SIRT versus LEN alone for patients with TACE-refractory HCC.

78 patients (39 in each arm) with TACE-refractory HCC will be enrolled in this study. The patients will receive either LEN+SIRT or LEN.

Lenvatinib (body weight ≥ 60 kg, 12mg P.O. QD; body weight < 60 kg, 8mg P.O. QD) will be administered to the patients and last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. For patients in the LEN+SIRT arm, lenvatinib will be started at 3-7 days after SIRT.

The primary end point of this study is objective response rate (ORR). The secondary endpoints are disease control rate (DCR), progression-free survival (PFS), time to response (TTR), duration of response (DOR), overall survival (OS), and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed or clinically diagnosed HCC
* Diagnosis of HCC with TACE refractoriness according to the criteria proposed by Japan Society of Hepatology (2021)
* Patients who have Tumor recurrence after surgical resection or ablation are allowed to be included
* At least one measurable intrahepatic target lesion
* Child-Pugh class A/B
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Tumor extent <70% liver occupation
* Candidates for SIRT must be confirmed suitable for SIRT after evaluation (including SPECT/CT evaluation after arterial perfusion with 99Tc-MAA)
* Adequate organ and hematologic function with platelet count ≥50×10^9/L, leukocyte >3.0×10^9/L, Neutrophil count ≥1.5×10^9/L, haemoglobin ≥85 g/L, ALT and AST≤5×ULN, albumin ≥28 g/L, total bilirubin ≤3× ULN, creatinine≤1.5×ULN, and prolongation of prothrombin time ≤4 seconds
* Life expectancy of at least 3 months

Exclusion Criteria:

* Extrahepatic metastasis
* Tumor thrombus involving main portal vein or both the first left and right branches of portal vein
* Vena cava invasion
* Patients who received prior hepatic arterial infusion chemotherapy (HAIC), radiotherapy, or systemic therapy, for HCC
* History of organ and cell transplantation
* History of esophageal or gastric variceal bleeding
* History of hepatic encephalopathy
* History of other malignancies
* Human immunodeficiency virus infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 years
  The percentage of patients who had a best overall tumor response rating of complete response (CR) or partial response (PR) according to mRECIST

SECONDARY OUTCOMES:
Disease control rate (DCR) | 3 years
  The percentage of patients who had a tumor response rating of CR, PR, or stable disease (SD) according to mRECIST.
Progression free survival (PFS) | 3 years
  The time from initiation of treatment until the first occurrence of disease progression or death from any cause, whichever occurs first.
Time to response (TTR) | 3 years
  The time from treatment initiation to first tumour remission (mRECIST)
Duration of response (DOR) | 3 years.
  Time from first tumor response to first disease progression (mRECIST) or death from any cause (whichever occurs first)
Overall survival (OS) | 4 years.
  The time from date of treatment initiation to death due to any cause
Adverse Events (AEs) | 3 years.
  Number of patients with AEs assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Mingyue Cai, Dr., Study Chair — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No